CLINICAL TRIAL: NCT00963833
Title: Study Evaluating Betaferons® Safety and Tolerability In Pediatric Patients With Multiple Sclerosis
Brief Title: Study Evaluating Betaferons Safety and Tolerability In Pediatric Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14438; BF0802 (Other: NIS Trial Alias)
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Non-interventional
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Patients under daily life treatment receiving Betaferon according to local product information.

SUMMARY:
Multiple Sclerosis (MS) is mainly known as a disease of young to middle adulthood but approximately 5% of all MS cases worldwide involve children that are younger than 16 years.

The aim of care of children with Multiple Sclerosis is to prevent or at least to delay any neurological and cognitive impairment as well as progression of the disease as far as possible. Therefore, it is very crucial to diagnose the disease at an early stage as immunomodulatory treatments are available that can delay the progression of Multiple SclerosisTreatment with the immunomodulatory agent Betaferon® in children diagnosed with RRMS and being 12 years or older has been approved by the health authorities. The aim of this observational study is to obtain further data on the safety, tolerability, and effectiveness of Betaferon® under daily living conditions.

As this is a non-interventional observational study, routine clinical practice is observed. The application of diagnostic measures and medications as well as physician visits follow the normal routine and is decided upon by the treating physician under recognition of the package insert.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive children and adolescents of 12 to 16 years of age at inclusion with a diagnosis of RRMS according to revised McDonald or Poser criteria and decision taken by the investigator to treat with Betaferon. The local Betaferon product information must be considered.

Exclusion Criteria:

* Contraindications stated in the local Betaferon product information; warnings and precautions must be considered.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Treatment naive children and adolescents aged 12 to 16 years at inclusion diagnosed with RRMS.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2009-12-17 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Betaferon in this patient population | Up 24 months

SECONDARY OUTCOMES:
Proportion of patients being relapse free | Up to 24 months
Time to first relapse | Up to 24 months
Annualized relapse rate | Up to 24 months
Disability progression measured by the expanded disability status scale (EDSS) | Up to 24 months
Outcome on neurological function | Up to 24 months
  e.g. IQ assessment using Standard Progressive Matrices (SPM) and Wechsler intelligence scale for children-fourth edition (WISCIV®), assessment of visual and motor integration using Beery VMI , and assessment of attention and concentration using d2 test.
Fatigue assessed by Fatigue Severity Scale (FSS) | Up to 24 months
MRI measurements (if available) | Up to 24 months
  e.g. number of new T2 lesions, number of new contrast enhancing lesions
MRI measurements and potential correlation with neuropsychological impairment | Up to 24 months
Laboratory outcomes | Up to 24 months
  Laboratory examinations: hemoglobin, mean corpuscular volume, platelets, leukocytes, ALAT/GPT, ASAT/GOT, Alkaline phosphatase, and Gamma-GT

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Many Locations, Austria
- Many Locations, Belgium
- Many Locations, Finland
- Many Locations, Germany
- Many Locations, Israel
- Many Locations, United Kingdom